CLINICAL TRIAL: NCT07286838
Title: Effects of Ciwujia Capsules/Compound Ciwujia Granules in the Treatment of Insomnia: a Multicenter, Prospective Real-world Study
Brief Title: Ciwujia Capsules/Compound Ciwujia Granules in the Treatment of Insomnia
Status: Not yet recruiting | Type: Observational
Sponsor: Hui Zhu (Other)
Collaborators: Huazhong University of Science and Technology (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Hui Zhu, Clinical Professor, Hubei Hospital of Traditional Chinese Medicine
Organization: Hubei Hospital of Traditional Chinese Medicine (Other)
Other Study IDs: HBZY2024-C62-02
Record Dates: First submitted 2025-11-20; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Insomnia Disorders
Keywords: Ciwujia Capsules/Compound Ciwujia Granules; Insomnia; real-world study
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Siberian ginseng root

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- insomnia patients
  Interventions: Drug: Ciwujia Capsules/Compound Ciwujia Granules

INTERVENTIONS:
Drug: Ciwujia Capsules/Compound Ciwujia Granules — Ciwujia Capsule may promote sleep because it has the function of strengthening the spleen, tonifying the kidney, and calming the mind.

SUMMARY:
The goal of this real-world study is to investigate the efficacy and safety of "Ciwujia Capsules/Compound Ciwujia Granules" in the treatment of insomnia in the clinical real-world. A total of 40000 patients with insomnia are assigned to 8 weeks of Ciwujia Capsules/Compound Ciwujia Granules treatment. The main question it aims to answer is:

1. Is there any significant reduction in Pittsburgh Sleep Quality Index (PSQI) score, Insomnia Severity Index (ISI) score, subjective sleep latency, sedatives or hypnotics use, and improvement in sleep maintenance after 8 weeks treatment of Ciwujia Capsules/Compound Ciwujia Granules?
2. Is Ciwujia Capsules/Compound Ciwujia Granules" a safe method for treating insomnia in adults?

DETAILED DESCRIPTION:
The investigators aimed to investigate the efficacy and safety of "Ciwujia Capsules/Compound Ciwujia Granules" in the treatment of insomnia in the clinical real-world. Eligible participants were adults aged 18-75 years old who had insomnia disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition [DSM5]), or self-reported history of disturbed sleep. The exclusion criteria were (1) self-reported allergy symptoms to any of the ingredients; (2) serious physical sickness; (3) a history of suicidal ideation or attempt, acute or chronic psychiatric condition not controlled by therapy; (4) baseline HAMD-17 score ≥17 or HAMA-14 score ≥14;(5) pregnant women; (6) history of drugs or alcohol abuse/dependence; (7) presence of other sleep disorders including sleep apnoea, restless legs syndrome; (8) participation in concurrent clinical trials.The primary outcome was the Pittsburgh Sleep Quality Index (PSQI) score. The secondary outcomes were the Insomnia Severity Index (ISI) score, sleep diary, sedatives or hypnotics usage, as well as the occurrence of adverse events at 8 weeks. The main question it aims to answer is:

1. Is there any significant reduction in Pittsburgh Sleep Quality Index (PSQI) score, Insomnia Severity Index (ISI) score, subjective sleep latency, sedatives or hypnotics use, and improvement in sleep maintenance after 8 weeks treatment of Ciwujia Capsules/Compound Ciwujia Granules?
2. Is Ciwujia Capsules/Compound Ciwujia Granules" a safe method for treating insomnia in adults?

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18-75 years old who had insomnia disorder (according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition [DSM5]), or self-reported history of disturbed sleep.

Exclusion Criteria:

* (1) self-reported allergy symptoms to any of the ingredients; (2) serious physical sickness; (3) a history of suicidal ideation or attempt, acute or chronic psychiatric condition not controlled by therapy; (4) baseline HAMD-17 score ≥17 or HAMA-14 score ≥14;(5) pregnant women; (6) history of drugs or alcohol abuse/dependence; (7) presence of other sleep disorders including sleep apnoea, restless legs syndrome; (8) participation in concurrent clinical trials.The primary outcome was the Pittsburgh Sleep Quality Index (PSQI) score.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 40000 patients with insomnia were included in this real-world study. Participants were adults aged 18-75 years old who had insomnia disorder, or self-reported history of disturbed sleep.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) score | From enrollment to the end of treatment at 8 weeks
  0-21, and higher scores mean a poorer sleep quality

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) score | From enrollment to the end of treatment at 8 weeks
  0-28, and higher scores mean a worse sleep problem
occurrence of adverse events | From enrollment to the end of treatment at 8 weeks

OTHER OUTCOMES:
Sleep diary | From enrollment to the end of treatment at 8 weeks
  providing daily information on subjective sleep onset latency, subjective total sleep time, subjective sleep quality, subjective wake after sleep onset, and subjective number of awakenings.
Sedatives or hypnotics use | From enrollment to the end of treatment at 8 weeks
  If it exists, provide information on the use of sedatives or hypnotics (e.g. drug names, dose, and duration)

IPD SHARING:
Plan to Share IPD: No